CLINICAL TRIAL: NCT04529499
Title: A Multi-center, Randomized, Double Blind, Placebo Controlled Clinical Trial Evaluating the Efficacy and Safety of Favipiravir in Moderate to Severe COVID-19 Patients
Brief Title: Clinical Trial Evaluating the Efficacy and Safety of Favipiravir in Moderate to Severe COVID-19 Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study met pre-defined criteria for futility at interim analysis
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVD-04-CD-001
Record Dates: First submitted 2020-08-19; First posted 2020-08-27 (Actual); Results first posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Covid19
Keywords: AVIGAN; Favipiravir; COVID-19; Phase 3
MeSH Terms: conditions — COVID-19 | interventions — favipiravir

STUDY DESIGN:
Intervention Model Description: 780 patients are randomized into two treatment groups at a 1:1 ratio, so as to have approximately 390 patients in favipiravir + supportive care group and 390 patients in placebo + supportive care group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a prospective, interventional, multi-centre, phase III, randomized, double blind, placebo-controlled, parallel design trial to evaluate the efficacy, safety and tolerability of favipiravir as adjunct ('add on') to supportive care, in comparison to placebo with supportive care, in the acute treatment of patients who have tested positive for SARS-CoV-2 and presenting with moderate to severe COVID-19.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- favipiravir + supportive care (Experimental): Frequency: Twice daily (morning and evening) Dosage Form: Tablets. Tablet Strength 200 mg. Dosage: 1,800 mg BID on Day 1 + 800 mg BID for next 9 days (maximum). On Day 1, the second dose will be administered with at least a 4-hour interval from administration of the first dose.
  Interventions: Drug: AVIGAN
- Placebo with Standard of Care (Placebo Comparator): Frequency: Twice daily (morning and evening) Dosage Form: Tablets Dosage: 9 tablets for BID on Day 1 + 4 tablets BID for next 9 days (maximum). On Day 1, the second dose will be administered with at least a 4-hour interval from administration of the first dose.
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: AVIGAN — Patients will be randomized to the favipiravir + supportive care group in a 1:1 ratio
  Other Names: Favipiravir
  Arms: favipiravir + supportive care
Drug: Placebo Comparator — Patients will be randomized to the placebo + supportive care group in a 1:1 ratio
  Other Names: Placebo
  Arms: Placebo with Standard of Care

SUMMARY:
This is a prospective, interventional, multi-centre, phase III, randomized, double blind, placebo-controlled, parallel design trial to evaluate the efficacy, safety and tolerability of favipiravir as adjunct ('add on') to supportive care, in comparison to placebo with supportive care, in the acute treatment of patients who have tested positive for SARS-CoV-2 and presenting with moderate to severe COVID-19.

This study will be conducted in two parts; Stage I - Main study and Stage II - Extended Follow up.

DETAILED DESCRIPTION:
Stage I - Main Study:

All the eligible patients will be randomized to receive either favipiravir + supportive care or placebo + supportive care. The treatment duration with the IMP will be for a period of 10 consecutive days. If the patient is discharged before Day 10, the patient will be required to continue the remainder of the treatment course of the assigned IMP at home. Patients in both the groups will receive supportive care, as appropriate. The duration of supportive care will be based upon Investigator's judgement and as per individual patient's requirement. The study data collection period will be up to 28 (+2) days.

Day 10 will be considered as the End of treatment (EOT) assessment.

1. If the patient remains in the hospital until Day 10, the EOT will be performed at the site and all the scheduled assessments for Day 10 will be performed
2. If the patient is discharged before Day 10, the EOT can be performed either as an onsite visit or will be performed at the patient's home :

   1. On-site visit: If the patient is able to visit the hospital on Day 10, procedures for an unscheduled visit will be performed.

      OR
   2. At home: If the patient is unable to visit the hospital for the EOT, study nurse or phlebotomist will visit the patient at his/her residence to collect blood sample for safety assessments. A telephonic follow up will be performed to enquire on treatment emergent AEs experienced, concomitant medication and COVID-19 associated symptom for assessment of clinical relapse.

Day 28 will be considered the end of study visit. If patient is discharged from the hospital before Day 28, the assessments mentioned in the end of study visit (Day 28) will be performed before the patient is discharged. After discharge, telephonic follow up will be performed on Day 10 (applicable only for patients who are discharged earlier than Day 10 and if patients are unable to visit the site for EOT on Day 10), Day 14, Day 21 and Day 28. The telephonic follow up will be as applicable for the individual patient, depending upon the actual day when (s)he is discharged. A 2-day window period is allowed for telephonic follow up.

In case the patient remains admitted in the hospital beyond Study Day 28, the end of study assessments will be performed for the patient on Day 28 (+2) days.

Stage I of the study will be completed when the 'Day 28' assessment is completed either as an in-patient assessment if the patient is still hospitalized, or as a telephonic follow up assessment if the patients are discharged earlier to Day 28.

Once all the patients complete the Stage I of the study, the database would be locked, and analysis will be performed.

Stage II - Extended Follow Up:

All the patients will be followed up for AEs or for 'clinical relapse' of COVID 19. Two telephonic follow up assessments will be performed on Day 42 and Day 60. An additional visit to the hospital (for further assessment) may be scheduled for such patients, if required.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 21 to 80 years (both inclusive)
2. Patients who have tested positive for SARS-CoV-2 by Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR) assay using a respiratory tract sample (either nasopharyngeal swab OR oropharyngeal swab OR nasal aspirate OR tracheobronchial aspirate) collected within 72 hours of randomization
3. Patients should be hospitalized
4. Patients having moderate or severe COVID-19* with a score of > 4 on the 10-point ordinal scale of clinical status used by WHO in the SOLIDARITY trial at baseline assessment [i.e., patients with blood oxygen saturation (SpO2) <95% at rest on room air at sea level and requiring supplemental oxygen].

   *Note: This includes patients clinically assigned as:

   I. 'moderate' COVID-19
   1. symptoms which could include fever, cough, sore throat, malaise, headache, muscle pain, gastrointestinal symptoms or shortness of breath with exertion and/or clinical signs, such as respiratory rate ≥20 breaths per minute or heart rate ≥90 beats per minute AND
   2. blood oxygen saturation (SpO2) of 94% at rest on room air at sea level

   II. 'severe' COVID-19
   1. symptoms which could include any symptom of moderate illness or shortness of breath at rest, or respiratory distress and/or clinical signs, such as respiratory rate ≥30 per minute or heart rate ≥125 per minute AND
   2. blood oxygen saturation (SpO2) ≤93% on room air at sea level or PaO2/FiO2 <300*

   The above-mentioned definitions of COVID-19 severity are adapted from the FDA Guidance document "COVID-19: Developing Drugs and Biological Products for Treatment or Prevention - Guidance for Industry Final Document" dated May 2020.
5. Female patients of childbearing potential*

   1. must have a negative serum pregnancy test at screening
   2. should not be lactating; and not planning to become pregnant/breast feed during the treatment period and for 7 days after the last dose of study medication.
   3. should commit to the use of TWO forms of study-acceptable contraception methods, including a barrier method (eg. diaphragm) along with one or more of the following methods of contraception for the duration of the treatment period and for 7 days after the last dose of study medication: i) hormonal methods [insertable, injectable, transdermal, or combination oral (estrogen+ progestin)], or ii) intrauterine contraceptive device

   Note: Female patients who are sexually abstinent or whose male sexual partner has undergone vasectomy at least three months prior to the start of study treatment in the trial may be enrolled at the Investigator's discretion, provided that they are counseled to remain sexually inactive for the duration of the study and understand the possible risks involved in getting pregnant during the study. Patients must also agree to use TWO forms of study-acceptable contraception methods should they become sexually active during the treatment period and for 7 days after the last dose of study medication.

   *Note: A female patient is considered of childbearing potential unless she is:
   1. postmenopausal for at least 12 months prior to study product administration, or
   2. without a uterus and/or both ovaries or has been surgically sterilized (i.e, tubal ligation or has a fallopian tube blocking coil) for at least 6 months prior to study product administration.
6. Male patients should agree to abstain from sexual intercourse or to use double-barrier contraception (e.g. condom with spermicide) for the duration of the treatment period in the study and for at least 7 days after receiving the last dose of study medication. Male patients should also avoid semen donation or providing semen for in-vitro fertilization during the above-mentioned duration.
7. Able and willing to provide informed consent
8. Able to understand the trial requirements and comply with trial medications and assessments in the opinion of the Investigator
9. Should not have received investigational treatment from participation in another clinical trial within 30 days prior to randomization in the current trial and agrees not to participate in other clinical studies during the entire study period

Exclusion Criteria:

1. Critically ill patients, defined as those who are candidates for endotracheal intubation and mechanical ventilation, oxygen delivered by high- flow nasal cannula, (heated, humidified, oxygen delivered via reinforced nasal cannula at flow rates >20 L/min with fraction of delivered oxygen ≥0.5), non-invasive positive pressure ventilation, Extracorporeal Membrane Oxygenation (ECMO) , or clinical diagnosis of respiratory failure (i.e., clinical need for one of the preceding therapies, but preceding therapies not able to be administered in setting of resource limitation) and those with shock (defined by systolic blood pressure (BP) <90 mm Hg, or diastolic BP <60 mm Hg or requiring vasopressors) or multi-organ dysfunction/failure, at baseline

   Note: The above-mentioned definition of 'critically ill' COVID-19 patients is as defined in the FDA Guidance document "COVID-19: Developing Drugs and Biological Products for Treatment or Prevention - Guidance for Industry Final Document" dated May 2020
2. Patients in whom the first onset of symptoms/signs suggestive of COVID-19 illness was observed >10 days earlier to the baseline assessment and randomization
3. Patients who have used interferon beta 1-a (IFN-β-1a) preparations or drugs with reported anti-viral action against SARS-CoV-2 (hydroxychloroquine sulfate, chloroquine phosphate, lopinavir-ritonavir combination drugs, ciclesonide, nafamostat mesylate, camostat mesylate) within 8 days after development of fever (≥37.5°C)

   Note: The above-mentioned exclusion criterion is not applicable in case of patients with history of human immunodeficiency virus infection or infective hepatitis in whom use of anti-viral drugs or interferons are prescribed for treatment of the underlying condition and who are currently receiving one or more of these medications (as maintenance treatment) at the time of randomization. The infection episode in question is a relapse of, or reinfection with SARS-CoV-2
4. Patients suspected to have a complication of congestive cardiac failure based on Investigator's clinical judgement
5. Patients with moderate and severe hepatic dysfunction equivalent to Grade B and Grade C in the Child-Pugh classification respectively
6. Patients with alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels > 5 times upper limit of normal (ULN) at screening evaluation
7. Patients with renal impairment requiring dialysis
8. Patients with serum uric acid higher than the ULN at screening evaluation
9. Patients with history of hereditary xanthinuria
10. Patients who have been diagnosed with xanthine urinary calculus
11. Patients with a history of gout or patients who are currently being treated for gout
12. Patients who are taking immunosuppressants
13. Patients who were administered Favipiravir in the past 30 days
14. Patients with known hypersensitivity reaction to Favipiravir

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2020-08-22 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sagar Munjal, MD, MS, Study Director — Dr Reddy's Laboratories, Inc
Locations (2):
- Kuwait (2):
  - Jaber Al-Ahmad Al-Sabah Hospital (South Surra), Kuwait City
  - Mishref Field Hospital (Mishref), Kuwait City

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period 22 AUG 2020 to 31 DEC 2020. The study was conducted at three hospitals in Kuwait ([Jaber Al Ahmad Al Jaber Al Sabah Hospital, Kuwait Mishref Field Hospital [(both of which are designated COVID-19 centers in Kuwait]) and Farwaniya Hospital, Kuwait)
Groups:
- Placebo + Supportive Care: Frequency: Twice daily (morning and evening) Dosage Form: Tablets Dosage: 9 tablets for BID on Day 1 + 4 tablets BID for next 9 days (maximum). On Day 1, the second dose will be administered with at least a 4-hour interval from administration of the first dose.
  Placebo Comparator: Patients will be randomized to the placebo + supportive care group in a 1:1 ratio
Period: Overall Study
Arm/Group | Favipiravir + Supportive Care | Placebo + Supportive Care
Started | 175 | 178
Discharged From Hospital Before Day 28 (Stage I) | 136 | 136
Completed 10-day Treatment Course of IMP (Stage I) | 150 | 147
Completed Day 14 Telephonic Visit (Stage I) | 107 | 102
Completed Day 21 Telephonic Visit (Stage I) | 119 | 120
Completed Day 28 Telephonic Visit (Stage I) | 134 | 131
Completed Days 14, 21 and 28 Telephonic Visits in Stage I (Stage I) | 98 | 94
Continue to be in Hospital as of Day 28 | 6 | 4
Completed Day 42 Telephonic Visit (Stage II) | 136 | 135
Completed Day 60 Telephonic Visit (Stage II) | 129 | 132
Completed Days 42 and 60 Telephonic Visits in Stage II (Stage II) | 126 | 130
Continued to be in Hospital When Study Was Terminated | 11 | 17
Completed (Stage I) | 139 | 138
Not Completed | 36 | 40
Not completed — Withdrawal by Subject | 9 | 11
Not completed — Physician Decision | 1 | 2
Not completed — Adverse Event | 4 | 4
Not completed — Death | 14 | 11
Not completed — Lost to Follow-up | 1 | 1
Not completed — Others | 7 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Favipiravir + Supportive Care | Placebo + Supportive Care | Total
Number analyzed (Participants) | 175 | 178 | 353
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (12.5) | 52.1 (12.5) | 51.9 (12.5)
Age, Customized [Count of Participants; unit: Participants]
  < 50 years | 70 | 74 | 144
  >/= 50 years | 105 | 104 | 209
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 58 | 115
  Male | 118 | 120 | 238
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 37 | 37 | 74
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 137 | 140 | 277
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Nationality of the subject ( as reported by subject)
  Participants
    Nationality: Bangladeshi | 5 | 7 | 12
    Nationality: Egyptian | 10 | 13 | 23
    Nationality: Indian | 15 | 20 | 35
    Nationality: Iranian | 2 | 6 | 8
    Nationality: Kuwaiti | 116 | 116 | 232
    Nationality: Filipino | 6 | 1 | 7
    Nationality: Others | 21 | 15 | 36
Body Mass Index [Mean (Standard Deviation); unit: kg / m^2] | 30.499 (6.351) | 31.042 (6.488) | 30.773 (6.416)
RT-PCR outcome at hospital admission [Count of Participants; unit: Participants]
  Positive on RT-PCR | 175 | 176 | 351
  Data Missing | 0 | 2 | 2
Clinical Status Score on WHO 10-point ordinal scale [Count of Participants; unit: Participants] — Clinical Severity of COVID-19 in subject was graded using WHO 10-point ordinal scale of clinical status ,where score 0 = "uninfected, no viral RNA" and score 10 = "death". Higher the scores more severe the disease ; increase in score (over baseline/ previous assessment) represents disease progression.
  Participants
    4 = Hospitalized, no oxygen therapy | 18 | 20 | 38
    5= Hospitalized, on oxygen | 156 | 156 | 312
    6 = Hospitalized, Oxygen by NIV or high flow | 1 | 1 | 2
    7= Mechanical Ventilation , p/f > 150 or s/f > 200 | 0 | 1 | 1
Baseline NEWS-2 score based clinical risk category [Count of Participants; unit: Participants]
  Low (NEWS 2 score: 0-4) | 86 | 96 | 182
  Low-Medium (NEWS 2 score of 3 in any individual parameter) | 0 | 1 | 1
  Medium (NEWS-2 Score: 5-6) | 74 | 69 | 143
  High (NEWS-2 score: >/= 7) | 14 | 10 | 24
  Data missing | 1 | 2 | 3
Randomization Strata to which assigned [Count of Participants; unit: Participants] — Subjects were assigned to strata of "moderate' or "severe" based on the disease severity category definitions in the FDA Guidance document COVID-19: Developing Drugs and Biological Products for Treatment or Prevention - Guidance for Industry Final Document dated May 2020
  Participants
    Moderate | 127 | 129 | 256
    Severe | 48 | 49 | 97
No. of days since onset of first symptom associated with COVID-19 [Median (Inter-Quartile Range); unit: days] — The time since onset of first COVID-19 symptoms is as reported by subject at time of enrollment
  days | 7.0 [5.0 to 7.0] | 7.0 [5.0 to 7.0] | 7.0 [5.0 to 7.0]

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Endpoint: Time to Resolution of Hypoxia (Stage I)
Description: This endpoint will be considered to have been met when the patient has attained a score of 4 or lower on the 10-point ordinal scale of clinical status used by WHO in the SOLIDARITY trial (maintaining a blood oxygen saturation of ≥ 95% at rest on room air at sea level) when evaluated over a period of 24 hours.
Time Frame: 1-28 days
Population: Analysis population (Intent-to-treat) was all randomized patients who had a clinical status score >4 on WHO 10-point ordinal scale at baseline
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Favipiravir + Supportive Care | Placebo + Supportive Care
Number analyzed (Participants) | 157 | 158
days | 7 [4 to 11] | 8 [5 to 12]
Statistical Analysis 1: Comparison: Favipiravir + Supportive Care vs Placebo + Supportive Care; Test type: Superiority; p = 0.67, Log Rank
Statistical Analysis 2: Comparison: Favipiravir + Supportive Care vs Placebo + Supportive Care; Test type: Superiority; Cox Proportional Hazard = 0.991, 95% CI 2-sided [0.767 to 1.280] — Favipiravir + supportive care in numerator and Placebo+ Supportive care in denominator for CPH ratio analysis

2. Secondary Outcome: Percentage of Patients Dying (All Cause (Stage I)
Description: Percentage of Patients dying from any cause over an assessment period from randomization until Day 28 or discharge from hospital (if discharge happens earlier)
Time Frame: 1-28 days
Population: Intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Favipiravir + Supportive Care | Placebo + Supportive Care
Number analyzed (Participants) | 175 | 178
Participants | 11 | 7
Statistical Analysis 1: Comparison: Favipiravir + Supportive Care vs Placebo + Supportive Care; Test type: Superiority; p = 0.34, Fisher Exact

ADVERSE EVENTS:
Time Frame: Baseline ( Day 1) to Day 28 or discharge or study discontinuation ( whichever was earlier)
Description: The All-Cause Mortality is reported for the population of randomized subjects ( = 'Intent-to-treat' population of the study) - 175 subjects in Favipiravir + supportive care and 178 subjects in placebo groups. Serious Adverse Events and Other (Not Including Serious) Adverse Events are reported for the safety population of the study (= randomized and received at least one dose of the study medication) - 168 subjects in Favipiravir + supportive care and 166 subjects in placebo groups.
Arm/Group | Favipiravir + Supportive Care | Placebo + Supportive Care
All-Cause Mortality (participants affected / at risk) | 14/175 | 11/178
Serious Adverse Events (participants affected / at risk) | 19/168 | 14/166
Other Adverse Events (participants affected / at risk) | 18/168 | 11/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Favipiravir + Supportive Care (N=168) | Placebo + Supportive Care (N=166)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1
Renal Impairment (Renal and urinary disorders) | 1 | 0
Hepatic Enzymes Increased (Investigations) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 1
Chest Pain (General disorders) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Favipiravir + Supportive Care (N=168) | Placebo + Supportive Care (N=166)
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 1
Blood uric acid increased (Investigations) | 1 | 1
Hemoglobin decreased (Investigations) | 1 | 0
Hepatic Enzymes Increased (Investigations) | 5 | 5
Lipids abnormal (Investigations) | 0 | 1
Liver function test increased (Investigations) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperuricemia (Investigations) | 8 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication will be a joint effort between Sponsors and Principal Investigator

DOCUMENTS (2):
  • Study Protocol (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/99/NCT04529499/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/99/NCT04529499/SAP_001.pdf